CLINICAL TRIAL: NCT06355570
Title: The Use of Auditory-visual Stimulation to Reduce Delirium Rates in Intensive Care Patients Post-cardiac Surgery: a Feasibility Study
Brief Title: Delirium After Cardiac Surgery in Intensive Care Units
Acronym: DaCsi-ICU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 331314; RFPR2324_29 (Other Grant/Funding Number: Imperial Health Charity); 24/YH/0011 (Other: UK Health Research Authority (Research Ethics Committee))
Record Dates: First submitted 2024-03-14; First posted 2024-04-09 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Intensive Care Unit Delirium; Cardiac Surgery; Post Operative Delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Intervention Model Description: 12-patient participants will be submitted to the study intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient Arm (Experimental): 12 patients will be recruited pre-operatively and submitted to the study intervention
  Interventions: Other: Personal Pictures; Other: Family Videos; Other: Family Videos - Intervention as required

INTERVENTIONS:
Other: Personal Pictures — Digital photos will be shown continuously at the patient's bedside for 12 hours a day (between 8 am to 8 pm).
Other: Family Videos — Family-recorded videos will be played three times at specific hours of the day - 9 am, 2 pm and 7 pm - throughout patient stay in the ICU
Other: Family Videos - Intervention as required — The last video shown will be re-played upon patient request and/or if patients develop ICU delirium.

SUMMARY:
STUDY SUMMARY

STUDY DESIGN The study will be conducted over twelve months in the Cardiac Intensive Care Unit (ICU) at Hammersmith Hospital, Imperial College Healthcare NHS Trust (ICHT). This study is a mixed methods research design that includes the collection of data through qualitative interviews, quality-of-life questionnaires and patients' medical records.

AIMS

* Determine the incidence of ICU delirium in ICHT following cardiac surgery
* Explore the compliance of outcome measures that diagnose ICU delirium
* Implement a family-focused sensory stimulation programme in the ICU
* Evaluate its useability and potential impact on patients, families and ICU staff

STUDY POPULATION 30 study participants (12 patients, 12 family members/friends and 6 ICU nurses)

ELIGIBILITY Study eligibility criteria are specific for each care group (patients, family members/friends and ICU nurses).

DURATION 12 months at Hammersmith Hospital, ICHT

DETAILED DESCRIPTION:
DaCsi-ICU is a mixed methods research study including the collection of data from patient's medical notes, interviews and quality of life questionnaires following the study schedule of assessments. This study also involves the implementation of an auditory-visual sensory stimulation package in the cardiac ICU at ICHT to participants enrolled in the study.

Digital photos will be shown continuously at the patient's bedside (8am-8pm) after cardiac surgery and will always have reference to time and date. Additionally, videos will be played throughout the patient's stay in the ICU at least three times per day (timepoints: 9am, 2pm,7pm) and upon participant request. Videos will be also played when participants show signs of ICU delirium to reduce its incidence and improve overall health outcomes. Simultaneously, data from patients' medical records will be routinely collected by the research team (e.g., Confusion Assessment Method-ICU, Richmond Agitation Sedation Scale, etc.) to assess whether patients develop delirium during their stay in the ICU.

Interviews with patients and families/friends will be held on three different occasions. The first one will be on the same day as ICU discharge, the second interview will be on the day of hospital discharge and the third one will be carried out up to a month following hospital discharge during their clinical follow-up appointment. Where possible, family members/friends and patient interviews will be conducted together (dyadic interviewing), but the possibility of performing interviews separately will be given so that participants feel able to discuss opinions freely. Nurses' interviews will be held as a one-off and after they have provided direct care to participants who received the proposed intervention.

Each patient will be followed up daily on the wards and once at the monthly follow-up clinic after ICU discharge, where cognitive and emotional assessments will be performed to evaluate delirium outcomes. The research team will also collect relevant information from participants' medical notes if any complications post-ICU discharge arise during inpatient and follow-up stages.

ELIGIBILITY:
INCLUSION CRITERIA

Patients

* Female and male patients over the age of 18
* Participants speaking English language and having mental capacity to consent
* Suitable to undergoing cardiac surgery at ICHT.

Family Members/Friends

* Nominated by the participant.
* Be willing to record videos and participate in the study.

Healthcare professionals

- Critical Care Nurses that have provided direct care to at least one patient who received the study intervention

EXCLUSION CRITERIA

Patients

* Female and male patients under the age of 18
* Unable to consent to the study pre-operatively
* Significant hearing/visual impairment
* Participants with learning disabilities, pre-existing delirium, dementia or other significant underlying cognitive morbidity
* Moribund participants, likely to die in the next 24 hours
* Participants that do not speak English language

Family Members/Friends

* Refuse to consent or gain assent
* Significant hearing/visual impairment
* Family members/friends that do not speak English language

Healthcare professionals

* Critical care nurses that have not been involved in the implementation of the intervention
* Refuse to consent or gain assent
* Significant hearing/visual impairment and non-English speaking

WITHDRAWAL CRITERIA:

Participants

* No longer willing to participate after consent
* Personal consultee wishing to withdraw participants from the study
* Patients that the clinical and/or research team deem too distressed to continue participating in the study
* Patients who have lost the capacity to participate in the study after hospital discharge

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-20 (Estimated)

PRIMARY OUTCOMES:
Feasibility of implementing the study intervention | 12 months
  The investigators plan to implement a family-focused auditory-visual sensory stimulation intervention to reduce ICU delirium rates post-cardiac surgery. Feasibility will be assessed by exploring facilitator factors and challenges that may arise during the implementation of this intervention. These elements will be recorded on a study reflective log and further discussed within the study team.

SECONDARY OUTCOMES:
Practicalities of introducing the study intervention | 12 months
  The investigators intend to explore the practical aspects of implementing an innovative non-pharmacological intervention in cardiac surgical ICU. The investigators also aim to collect nursing checklists, routinely liaise with the local clinical/research team and explore any additional internal approvals to implement the study in the ICU.
Acceptability of implementing the study intervention | 12 months
  The investigators plan to conduct qualitative interviews with critical care staff, patients and family members/friends to explore their acceptance and experience of taking part in the study.
Short-term delirium outcomes post-ICU discharge | 12 months
  The investigators intend to conduct an extra qualitative interview with patients and family members/friends up to a month after hospital discharge to explore any post-ICU delirium complications. Additionally, cognitive and emotional questionnaires (The Mini-Mental State Examination, General Anxiety Disorder-7 and Patient Health Questionnaire-9) will be performed at two different time points to further explore post-ICU delirium outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Reguenga, BSN, Principal Investigator — Imperial College Healthcare NHS Trust
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] De Azinheira Reguenga MJ, Lampridou S, Pattison N, Brett SJ, Soni S. The use of audio-visual aids to reduce delirium after cardiac surgery in intensive care units (DaCSi-ICU): A feasibility study protocol. PLoS One. 2025 Apr 24;20(4):e0320935. doi: 10.1371/journal.pone.0320935. eCollection 2025. PMID 40273276